CLINICAL TRIAL: NCT02382952
Title: Pilot Study Differential Dissector™ for Blunt Dissection
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 14-2888
Record Dates: First submitted 2015-03-03; First posted 2015-03-09 (Estimated); Last update posted 2016-08-05 (Estimated); Status verified 2016-07

CONDITIONS: Surgical Adhesions; Blood Loss, Surgical
Keywords: Abdominal surgery; Pelvic surgery; Stoma takedown; Bowel resection; Lysis of abdominal adhesions
MeSH Terms: conditions — Tissue Adhesions; Blood Loss, Surgical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Differential Dissector (Experimental): For patients in the study device group, blunt dissection will be performed with the Differential Dissector whenever the surgeon believes its use is appropriate.
  Interventions: Device: Differential Dissector
- Standard Dissection Method (Active Comparator): For patients in the control group, blunt dissection will be performed by standard method.
  Interventions: Other: Standard Dissection Method

INTERVENTIONS:
Device: Differential Dissector
  Arms: Differential Dissector
Other: Standard Dissection Method
  Arms: Standard Dissection Method

SUMMARY:
The primary purpose of this study is to evaluate the quality of blunt dissection during abdominal and pelvic surgery involving dissection of adhesions, separation of blood vessels and neurovascular structures while preserving the integrity of these structures.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18
* Patient will be undergoing open abdominal surgery
* Patient willing and able to provide his/her own consent

Exclusion Criteria:

* Current alcohol or other substance abuse
* Current incarceration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-03; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Operative Blood Loss | From start of surgery to wound closure
Post-operative Blood Loss | After surgical closure and drain insertion through drain removal

CONTACTS AND LOCATIONS:
Overall Officials: Mark Koruda, MD, Principal Investigator — University of North Carolina, Chapel Hill

IPD SHARING:
Plan to Share IPD: No